CLINICAL TRIAL: NCT04686071
Title: The Efficiency of the PNF Method in Assessing Functional Performance in Early Stage Patients Following Knee Arthroplasty
Brief Title: The Efficiency of the PNF Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Maicki, Principal, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNEE2018
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Knee Arthroplasty
Keywords: gonarthrosis, knee replacement, osteoarthritis, PNF method
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients were randomly divided into two groups which differed in the type of a 10-day treatment model used after the operation.Specifying the group was done by drawing a sealed, opaque envelope: an envelope with an even number ment PNF treatment, while an odd number ment traditional therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF method (Experimental)
  Interventions: Other: PNF method
- standard rehabilitation (Other)
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: PNF method — Treatment in the study group was conducted with PNF method with a use of indirect training based on irradiation phenomenon. The program included: proprioceptive stimulation of the operated limb, improving trunk stabilization and active control, active foot training, muscle strength facilitation of lower limbs in closed kinematic chain with considering periarticular stabilization within the operated knee joint as well as exercises improving mobility of the operated knee, verticalization and locomotion with emphasis on the stance phase.
  Arms: PNF method
Other: Standard rehabilitation — In the control group standard rehabilitation protocol was used in patients following TKA, which is mainly based on activities in open chains (passive exercises with continuous passive motion (CMP) device, active exercises, isometric, active resistance, patella mobilization, deep tissue massage, verticalization and gait relearning).
  Arms: standard rehabilitation

SUMMARY:
Background: Early rehabilitation following knee arthroplasty is an integral part of medical management which reduces the time of patient's stay at hospital and eliminates the risk of post-operative complications. The absence of consensus on the most efficient post-operative rehabilitation strategy and shortage of practices based on evidence lead to seek new therapeutic solutions. Therefore the goal of this study is to evaluate the efficiency of the PNF method in assessing functional performance in early stage patients following knee arthroplasty Material and methods: The study was conducted among 96 patients (66,34 years ±7,29) who were qualified to total knee arthroplasty. The patients were randomly divided into two groups. In the control group standard rehabilitation protocol was implemented while post-operative treatment in the study group based on PNF method. All the patients were tested on the day of admission to the hospital and after completing a 10-day rehabilitation program. Structural and functional parameters of the operated knee (muscle strength, range of motion, circuit measurements) as well as functional abilities (Staffelstein Score, Lequesne Index) were evaluated.

Key words: gonarthrosis, knee replacement, osteoarthritis, PNF method

DETAILED DESCRIPTION:
Involution changes of the human body are characteristics of aging. A decrease in physical activity as well as increased life expectancy can be a factor in the development of many pathological changes in the movement system resulting in increase in the number of people with diagnosed osteoarthritis (OA) [1]. Epidemiological studies indicate that osteoarthritis affects up to 40 million people in Europe [2], including 10% of men and 13% of women above 60 years of age with knee degenerative changes [3]. It is estimated that in Poland over 8 million people suffer from osteoarthritis, out of which 25% have gonarthrosis [4]. Osteoarthritis detracts from the quality of life and leads to malfunction and this is therefore necessary to early implement prevention and treatment actions which allow for keeping functional performance and protection against development of destructive changes [5].The study will be conducted in Cracow Rehabilitation and Orthopedics Centre. The study group will be qualified to the total knee arthroplasty due to pain caused by advanced knee osteoarthritis. . The patients will be randomly divided into two groups which differed in the type of a 10-day treatment model used after the operation.

In the control group standard rehabilitation protocol will be used in patients following TKA, which is mainly based on activities in open chains (passive exercises with continuous passive motion (CMP) device, active exercises, isometric, active resistance, patella mobilization, deep tissue massage, verticalization and gait relearning). Treatment in the study group will be conducted with PNF method with a use of indirect training based on irradiation phenomenon. The program included: proprioceptive stimulation of the operated limb, improving trunk stabilization and active control, active foot training, muscle strength facilitation of lower limbs in closed kinematic chain with considering periarticular stabilization within the operated knee joint as well as exercises improving mobility of the operated knee, verticalization and locomotion with emphasis on the stance phase.

In this study, an attempt will be made to analyze treatment effects on parameters assessing function of the knee joint and functional abilities in daily living with a use of a classic rehabilitation protocol and PNF method in patients following TKA. To evaluate efficacy of the therapy all the patients will be tested on the day of admission to the hospital and on the last day of the treatment. Structural and activity parameters of the operated knee joint will be evaluated, such as muscle strength (6-point Lovett scale), range of motion (digital inclinometer) and circuits measurement (centimeter). Circuits were measured on the level of the knee joint articular space, 10 cm (Thigh I) and 20 cm (Thigh II) above the articular space as well as on the level of lower leg (the widest point). Scales based on a subjective evaluation, such as Staffelstein Score and Lequesne Index will be performed to assess functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* the total knee arthroplasty due to pain caused by advanced knee osteoarthritis.

Exclusion Criteria:

* stroke

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
muscle strength test | baseline
  (6-point Lovett scale)
muscle strength test | at 10 days
  (6-point Lovett scale)
range of motiondigital inclinometer | baseline,
range of motiondigital inclinometer | at 10 days
circuits measurement (centimeter) | baseline, at 10 days
  Circuits were measured on the level of the knee joint articular space, 10 cm (Thigh I) and 20 cm (Thigh II) above the articular space as well as on the level of lower leg (the widest point).
Staffelstein Score | baseline,
  subjective evaluation to assess functional abilities
Lequesne Index | at 10 days
  subjective evaluationto assess functional abilities

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Krakowskie Centrum Rehabilitacji i Ortopedii, Krakow, Małopolska
  - Tomasz Maicki, Krakow

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: available
Access Criteria: on email request: tomasz.maicki@uj.edu.pl

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Conaghan PG, Kloppenburg M, Schett G, Bijlsma JW; EULAR osteoarthritis ad hoc committee. Osteoarthritis research priorities: a report from a EULAR ad hoc expert committee. Ann Rheum Dis. 2014 Aug;73(8):1442-5. doi: 10.1136/annrheumdis-2013-204660. Epub 2014 Mar 13. PMID 24625626
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Chojnacki M, Kwapisz A, Synder M, Szemraj J. [Osteoarthritis: etiology, risk factors, molecular mechanisms]. Postepy Hig Med Dosw (Online). 2014 Jan 2;68:640-52. doi: 10.5604/17322693.1103551. Polish. PMID 24864114
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] National Clinical Guideline Centre [editorial]. Osteoarhritis: care and management in adults. NICE 2014;177: 1-36
- [Background] Davila Castrodad IM, Recai TM, Abraham MM, Etcheson JI, Mohamed NS, Edalatpour A, Delanois RE. Rehabilitation protocols following total knee arthroplasty: a review of study designs and outcome measures. Ann Transl Med. 2019 Oct;7(Suppl 7):S255. doi: 10.21037/atm.2019.08.15. PMID 31728379
- [Background] Papalia R, Campi S, Vorini F, Zampogna B, Vasta S, Papalia G, Fossati C, Torre G, Denaro V. The Role of Physical Activity and Rehabilitation Following Hip and Knee Arthroplasty in the Elderly. J Clin Med. 2020 May 9;9(5):1401. doi: 10.3390/jcm9051401. PMID 32397459